CLINICAL TRIAL: NCT07389187
Title: An Open-Label, Single-Arm, Exploratory Study to Evaluate the Safety and Preliminary Efficacy of LC-K76 Plus Anti-PD-1 Therapy in Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: Safety and Preliminary Efficacy Evaluation of LC-K76 Plus Anti-PD-1 Therapy in Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Ren Shancheng, Professor, Chief of Urology, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LC-K76-201
Record Dates: First submitted 2025-12-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: mCRPC
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LC-K76 + Tislelizumab + ADT (Experimental): Participants receive oral LC-K76 combined with intravenous Anti-PD-1 monoclonal antibody (Tislelizumab) and standard androgen deprivation therapy (ADT). Treatment continues for 24 weeks.
  Interventions: Dietary Supplement: LC-K76; Drug: Tislelizumab; Drug: Standard Androgen Deprivation Therapy (ADT)

INTERVENTIONS:
Dietary Supplement: LC-K76 — Oral administration, 1.2 g twice daily (BID), taken 30 minutes before breakfast and dinner.
Drug: Tislelizumab — Intravenous infusion, 200 mg every 3 weeks (Q3W).
Drug: Standard Androgen Deprivation Therapy (ADT) — Maintenance of ADT using GnRH agonist or antagonist (e.g., Goserelin, Leuprorelin, Triptorelin, or Degarelix).

SUMMARY:
This open-label, single-arm study evaluates the safety and preliminary efficacy of LC-K76 combined with Tislelizumab and ADT in 10 patients with Metastatic Castration-Resistant Prostate Cancer (mCRPC) who progressed on prior therapies. Participants will receive oral LC-K76 and intravenous Tislelizumab for a 24-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged 18 to 85 years.
2. Histologically confirmed prostate adenocarcinoma, without small cell carcinoma components.
3. Metastatic Castration-Resistant Prostate Cancer (mCRPC) with disease progression after at least one novel endocrine therapy (e.g., abiraterone or enzalutamide) and/or docetaxel chemotherapy.
4. Evidence of bone metastasis on PSMA-PET-CT or bone scan (ECT).
5. Serum testosterone at castration levels (< 50 ng/dL or 1.75 nmol/L).
6. ECOG performance status ≤ 2.
7. Life expectancy > 6 months.
8. Adequate bone marrow, hepatic, and renal function.
9. Willing to undergo biopsies before and during treatment

Exclusion Criteria:

1. Lack of pathological evidence for prostate cancer.
2. Other primary malignant tumors active or requiring treatment within the past 3 years.
3. Has visceral metastases.
4. Poorly controlled diabetes after continuous insulin therapy.
5. Significant abnormalities in laboratory values at randomization (Hb < 90 g/L; Neutrophils < 1.5x10^9/L; Platelets < 75x10^9/L; ALT/AST > 2.5xULN; Bilirubin > 1.5xULN; eGFR < 60 mL/min/1.73m^2) .
6. Severe cardiopulmonary disease or high-risk conditions.
7. Prior therapy with any immune checkpoint inhibitors (e.g., anti-PD-1/PD-L1).
8. Intolerance to anti-PD-1 monoclonal antibody or dandelion extracts.
9. History of severe drug allergies.
10. Factors affecting drug intake/absorption (e.g., swallowing difficulty, chronic diarrhea).
11. Concurrent psychiatric or neurological conditions

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From baseline to primary completion, which may take up to 24 to 48 weeks
  The Incidence of Adverse Events is defined as the proportion of subjects in a clinical trial who experience at least one Adverse Event (AE) during the defined observation period, which is assessed by CTCAE 5.0.

SECONDARY OUTCOMES:
PSA Response Rate | From baseline to primary completion, which may take up to 24 to 48 weeks
Disease control rate (DCR) | From baseline to primary completion, which may take up to 24 to 48 weeks
  Defined as the proportion of subjects whose best overall response, assessed per RECIST 1.1 and PCWG3, is Complete Response (CR), Partial Response (PR), or Stable Disease (SD) .
Radiographic Progression-Free Survival (rPFS) | From baseline to primary completion, which may take up to 24 to 48 weeks
  Defined as the time from treatment initiation to the first objective evidence of disease progression as assessed by radiographic imaging, or death from any cause, whichever occurs first.
Time to First Skeletal-Related Event (SRE) | From baseline to primary completion, which may take up to 24 to 48 weeks
  Defined as the interval from the date of treatment initiation to the date of the first occurrence of any of the following clinically significant events attributable to bone metastasis: pathological fracture (vertebral or non-vertebral), palliative radiation therapy to bone for pain relief, surgical intervention to bone to prevent or treat a fracture or spinal cord compression, or confirmed spinal cord compression.

CONTACTS AND LOCATIONS:
Locations (1):
- Changzheng hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No